CLINICAL TRIAL: NCT00849030
Title: A Randomised, Double Blind Trial Comparing Arimidex Alone With Nolvadex Alone With Arimidex and Nolvadex in Combination, as Adjuvant Treatment in Post-Menopausal Women With Breast Cancer
Brief Title: ATAC - Arimidex, Tamoxifen Alone or in Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1033IL/0029; D5392C00029
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Arimidex 1mg + Nolvadex placebo
  Interventions: Drug: Anastozole (Arimidex); Drug: Tamoxifen (Nolvadex) placebo
- 2 (Active Comparator): Arimidex placebo + Nolvadex 20mg
  Interventions: Drug: Tamoxifen (Nolvadex); Drug: Anastozole (Arimidex) placebo
- 3 (Active Comparator): Arimidex 1mg + Nolvadex 20mg
  Interventions: Drug: Anastozole (Arimidex); Drug: Tamoxifen (Nolvadex)

INTERVENTIONS:
Drug: Anastozole (Arimidex) — 1mg, orally, once daily
  Other Names: Arimidex
  Arms: 1; 3
Drug: Tamoxifen (Nolvadex) — 20mg, orally, once daily
  Other Names: Nolvadex
  Arms: 2; 3
Drug: Anastozole (Arimidex) placebo — 1mg, orally, once daily
  Arms: 2
Drug: Tamoxifen (Nolvadex) placebo — 20mg, orally, once daily
  Arms: 1

SUMMARY:
The aim of this study is to test whether Arimidex alone or in combination with Tamoxifen is beneficial in the treatment of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven operable invasive breast cancer
* Patients who have completed all primary surgery and chemotherapy (if given), and are candidates to receive hormonal adjuvant therapy
* Women defined as post-menopausal

Exclusion Criteria:

* Patients in whom there is any clinical evidence of metastatic disease
* Patients who, for whatever reason (e.g. confusion, infirmity, alcoholism), are unlikely to comply with trial requirements
* Patients whose chemotherapy was started more than 8 weeks (ie 56 days) after completion of primary surgery or whose chemotherapy was completed more than 8 weeks (ie 56 days) before starting randomised treatment

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9358 (Actual)
Dates: Start 1996-07; Primary Completion 2001-06 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to recurrence of breast cancer | Earliest of local or distant recurrence, new primary breast cancer, or death
Safety and side effects | Earliest of local or distant recurrence, new primary breast cancer, or death

SECONDARY OUTCOMES:
Time to distant recurrence | Earliest of local or distant recurrence, new primary breast cancer, or death
Survival | Earliest of local or distant recurrence, new primary breast cancer, or death
New breast primaries | Earliest of local or distant recurrence, new primary breast cancer, or death